CLINICAL TRIAL: NCT03361891
Title: WalkMORE: Volunteer Walking Coach Program for Hospitalized Internal Medicine Patients, a Pilot Randomized Controlled Trial
Brief Title: WalkMORE: Volunteer Walking Coach Program for Hospitalized Internal Medicine Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ReDA 4304
Record Dates: First submitted 2017-11-27; First posted 2017-12-05 (Actual); Last update posted 2019-03-15 (Actual); Status verified 2019-03

CONDITIONS: Early Ambulation

STUDY DESIGN:
Intervention Model Description: Patients will be randomized via REDCap (Research Electronic Data Capture), a secure, centralized web-based randomization module to:
  1. Standard of care; or
  2. WalkMORE Ambulation program + Standard of care. Patients will ambulate with a trained WalkMORE Volunteer Coach two times per day; once in the morning (0900-1200hrs) and once in the afternoon (1300-1700hrs), Monday- Friday, until hospital discharge. Patients randomized to the WalkMORE intervention will be assessed daily by the Research Coordinator to ensure patients remain fit for independent ambulation. The duration of each walking session will be determined daily by the RC and the medical team.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Patients receive no intervention
- WalkMORE group (Experimental): WalkMORE Ambulation program. Patients will ambulate with a trained WalkMORE Volunteer Coach two times per day; once in the morning (0900-1200hrs) and once in the afternoon (1300-1700hrs), Monday- Friday, until hospital discharge.
  Interventions: Behavioral: WalkMORE Group

INTERVENTIONS:
Behavioral: WalkMORE Group — Hospitalized Internal Medicine patients will walk with trained volunteer coaches twice daily until hospital discharge
  Arms: WalkMORE group

SUMMARY:
Patients admitted to hospital typically experience periods of decreased activity or bed-rest. This reduced activity level leads to deconditioning - a loss of muscle mass, muscle strength (by 2-5% per day), and muscle shortening. Even among patients who were ambulatory at the time of admission, deconditioning has been linked with deleterious effects, such as increased rates of falls, functional decline, and frailty. Furthermore, it has been suggested that the physiological stresses associated with hospitalization - including deconditioning, as well as sleep deprivation and poor nutrition - makes discharged patients vulnerable to recurrent or new illnesses and to frailty. This physiological stress-induced vulnerability has been coined post-hospital syndrome and is thought to have a role in most hospital readmissions.

The investigators hypothesize that by engaging ambulatory patients to walk with trained volunteer coaches, patients will increase their amount of walking, have less deconditioning and functional decline, and consequently, fewer falls. Furthermore, the investigators anticipate that patients who walk with a trained coach will have reduced length-of-stay in hospital and decreased likelihood of readmission. Finally, as shown in other programs trialing health coaches, the investigators anticipate an overall improvement in the patient experience.

Our aim is to demonstrate the feasibility of an intentional walking protocol called WalkMORE, which pairs trained volunteer coaches with ambulatory patients admitted to the Internal Medicine unit (4th floor University Hospital), aimed at decreasing deconditioning through increased walking.

DETAILED DESCRIPTION:
WalkMORE is a single-center randomized controlled trial. The investigators will enroll up to 300 ambulatory patients admitted to the Internal Medicine unit (located on the 4th floor of University Hospital) who are >18 years of age and are anticipated to require a >48 hour hospital admission. A maximum of 6 patients will be assigned to each treatment arm at any given time. The investigators will recruit patients into the WalkMORE program over a 3-month period. The research coordinator (RC) will screen patients admitted to the Internal Medicine unit in the preceding 24-hour period to identify patients who fulfill the eligibility criteria. Patients will be randomized via REDCap (Research Electronic Data Capture), a secure, centralized web-based randomization module to:

1. Standard of care; or
2. WalkMORE Ambulation program + Standard of care. Patients will ambulate with a trained WalkMORE Volunteer Coach two times per day; once in the morning (0900-1200hrs) and once in the afternoon (1300-1700hrs), Monday- Friday, until hospital discharge. Patients randomized to the WalkMORE intervention will be assessed daily by the RC to ensure patients remain fit for independent ambulation. The duration of each walking session will be determined daily by the RC and the medical team.

After obtaining written informed consent from eligible patients the RC will randomize patients, collect demographics, hospital admission details and perform a quality of life survey (EQ-5D) with all patients. All patients will be assigned a scientific pedometer on the day of randomization. The modus Health StepWatch™ is an activity monitor worn on the ankle via a velcro strap. It is a small, lightweight device that will count and record patients' steps throughout their hospital stay. The device is smaller than a deck of cards (7.5 x 5.0 x 2.0 cm) and weighs 38 grams and will be installed by the RC. The total number of steps recorded on the pedometer will be collected for each patient every day until hospital discharge. For patients randomized to the WalkMORE intervention arm, the total number of minutes walked with a volunteer coach will also be recorded for each session until discharge. Functional ability will be measured on the third day post-randomization and every three days thereafter until hospital discharge, using the Timed Up and Go test (patients will be asked to stand up from a chair, walk three metres, turn around, walk back to the chair, and sit). After hospital discharge the RC will follow up with patients for 2 brief telephone interviews. On day 3 after discharge, Patient Satisfaction surveys will be conducted by the RC to assess patient satisfaction with their experience with the WalkMORE program. These telephone surveys will be reviewed and approved by Lisa Hawthorne of the Patient Experience Office. On day 30 after discharge the RC will contact patients to conduct a brief quality of life survey and to collect data regarding clinical outcomes (ER visits, re-hospitalizations, and falls). Each telephone interview is expected to last approximately 10-15 minutes.

ELIGIBILITY:
Inclusion Criteria:

1. Capable and appropriate for independent ambulation (with or without gait aids) as determined by the health care team at time of admission
2. Cognitively safe for participation
3. Anticipated to remain hospitalized ≥48 hours
4. Age >18 years

Exclusion Criteria:

1. Preexisting condition precludes patient from independent ambulation at time of admission.
2. Active medical condition precludes patient from safely participating.
3. Preexisting condition or active medical condition renders patient unfit to participate as judged by the admitting team.
4. Patients who refuse to participate or are unable to provide informed consent.
5. Patients that are non-English speaking.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2018-06-06 (Actual); Primary Completion 2018-12-10 (Actual); Study Completion 2019-01-09 (Actual)

PRIMARY OUTCOMES:
Patient Recruitment | 3 months
  Ability to recruit sufficient number of patients

SECONDARY OUTCOMES:
Patient Safety | 6 months
  Number of participants that experience a fall during the study intervention as reported by WalkMORE volunteer coaches.

CONTACTS AND LOCATIONS:
Locations (1):
- LHSC-University Hospital, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No